CLINICAL TRIAL: NCT03924661
Title: A Single Arm, Non-randomized, Multi-center Clinical Study of the SJM Masters HP 15mm Rotatable Mechanical Heart Valve as Aortic Valve Replacement Therapy
Brief Title: SJM Masters HP 15mm Rotatable Mechanical Heart Valve as Aortic Valve Replacement Therapy
Status: Active, not recruiting | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: ABT-CIP-10237
Record Dates: First submitted 2019-04-16; First posted 2019-04-23 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Aortic Valve Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Single Arm: Surgical treatment of a diseased, damaged, or malfunctioning aortic valve using SJM™ Masters Series Hemodynamic Plus (HP) 15mm aortic mechanical heart valve surgical replacement device
  Interventions: Device: Aortic Valve Replacement

INTERVENTIONS:
Device: Aortic Valve Replacement — SJM™ Masters Series Hemodynamic Plus (HP) 15mm aortic mechanical heart valve as a replacement device for patients with a diseased, damaged, or malfunctioning aortic valve

SUMMARY:
This PAS is an observational, non-randomized, multi-center, single arm, clinical study to evaluate long term safety and effectiveness of the SJM™ Masters Series Hemodynamic Plus (HP) 15mm aortic mechanical heart valve (15 AHPJ-505) as a replacement device for pediatric patients with a diseased, damaged, or malfunctioning aortic valve.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for prospectively enrolled subjects

  * Subject's legal guardian must provide written informed consent prior to any clinical study related procedure.
  * Subject requires aortic valve replacement and is intended to be implanted with a 15mm SJM15 AHPJ-505 MHV as determined by the implanting physician in accordance with the Instructions for Use.
  * The legal guardian and site agree to follow the subject per the assessment schedule and complete all required assessments per this protocol for the duration of the clinical study.
* Inclusion criteria for retrospectively enrolled subjects :

In an effort to ensure data on all real-world use conditions are consistently collected and reported on, a subject is eligible to participate in this post-approval study if he/she meets all of the following inclusion criteria and meets no exclusion criterion. For those subjects with a previous implant attempt to be eligible for study participation, the following inclusion criteria must be met:

* Echocardiography data at a time point greater than 90 days is available or may be acquired.
* An implant was attempted with the 15mm MHV, where implant attempt is defined as the device physically contacting the subject's cardiac anatomy.
* Either:
* For living subjects who already received the 15mm MHV, the legal guardian signs the study informed consent for this protocol allowing access to all relevant historical medical information, and complete all required assessments according to this protocol from the time of consent going forward (if applicable).

OR

* For subjects who are deceased or explanted, an implantation with 15mm MHV was attempted and the subject's legal guardian provides written informed consent for retrospective data collection of patient and study valve related information through death or explant of the study device.

Exclusion Criteria:

* Exclusion criteria for prospectively enrolled subjects:

Subject has a contraindication to anticoagulant/antiplatelet medication.

* Exclusion criteria of retrospectively enrolled subjects: None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This clinical study will enroll male and female subjects from the pediatric population. Subjects must meet all eligibility criteria and written and signed informed consent must be obtained from the subject's legal guardian prior to starting the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Rate of total serious valve-related adverse events | 5 Years
  actuarial (Kaplan-Meier) rate of total serious valve-related adverse events experienced through 5 years post implant or until the valve is removed/replaced. Valve-related adverse events to be evaluated are:
  * Death;
  * Endocarditis;
  * Hemorrhage (whether or not due to anticoagulant/antiplatelet medication);
  * Nonstructural dysfunction (including perivalvular leak, hemolysis, and hemolytic anemia);
  * Reoperation (including valve explant, not due to anatomical growth of the subject);
  * Structural valve deterioration;
  * Thromboembolism
  * Valvular thrombosis
Peak gradient as assessed by echocardiography | Up to 5 years
  Peak gradient as assessed by echocardiography at 30 Days, 6 Months, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year
Mean gradient as assessed by echocardiography | Up to 5 years
  Mean gradient as assessed by echocardiography at 30 Days, 6 Months, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year
Valvular regurgitation as assessed by echocardiography | Up to 5 years
  Valvular regurgitation as assessed by echocardiography at 30 Days, 6 Months, 1 Year, 2 Year, 3 Year, 4 Year, 5 Year

SECONDARY OUTCOMES:
Number of all-cause deaths | 1 Year
Number of valve-related deaths | 1 Year
Number of reoperations or explants excluding replacement due to somatic growth | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Abbott Medical Devices
Locations (13):
- United States (9):
  - Children's Hospital Los Angeles (USC), Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Sutter Medical Center, Sacramento, Sacramento, California
  - Variety Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Dell Children's Medical Center, Austin, Texas
  - Children's Medical Center Dallas, Dallas, Texas
- Germany (4):
  - Sana - Herzchirurgische Klinik Stuttgart GmbH, Stuttgart, Baden-Wurttemberg
  - Deutsches Herzzentrum München des Freistaates Bayern, München, Bavaria
  - Herzzentrum Leipzig GmbH, Leipzig, Saxony
  - Medizinische Hochschule Hannover, Hanover